CLINICAL TRIAL: NCT05909475
Title: Supplementation With GKEX Sports Probiotic Combo for Muscle Gain and Fat Loss Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, Chi-Chang Huang, Distinguished Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 22-022
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sport Nutrition; Probiotic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 2 caps daily use.
  Interventions: Other: Placebo
- GKEX (Experimental): GKEX group. Probiotic capsules contain 10 billion CFU (colony forming units) of GKEX, , 2 caps daily use.
  Interventions: Dietary Supplement: GKEX

INTERVENTIONS:
Dietary Supplement: GKEX — GKEX group. Probiotic capsules contain 10 billion CFU (colony forming units) of GKEX, , 2 caps daily use.
  Arms: GKEX
Other: Placebo — The placebo capsule contains microcrystalline cellulose, 2 caps daily use.
  Arms: Placebo

SUMMARY:
Objective: To discuss the "GKEX Sports Probiotics Combination (hereinafter referred to as GKEX)", a product commissioned by Grape King Biotechnology Co., Ltd., and its effects on increasing muscle mass, muscle strength, physical performance and improving body composition when combined with resistance exercise training. Method: The experiment adopts a double-blind design. After screening, 52 subjects (20 males and 32 females) were randomly divided into two groups, each with 10 males and 16 females: (1) placebo without GKEX probiotics Capsule group (Placebo) (2 capsules/day), (2) GKEX group (GKEX) (1x1010 CFU/capsule, 2 capsules/day). All subjects received daily supplementation samples for 6 weeks and received resistance exercise training three times a week. Before the intervention and 6 weeks after the intervention, the diet evaluation, systemic and resistive body composition, muscle ultrasound, muscle strength, maximum oxygen uptake, explosive power, anaerobic power, etc. were detected respectively.

ELIGIBILITY:
Inclusion Criteria:

* The tissues and organs of the body are functioning normally
* no disease, fatigue, or weakness
* independent and flexible activities

Exclusion Criteria:

* With a history of cardiovascular disease, hypertension, metabolic disease, asthma or cancer diagnosed by a physician
* BMI≧27
* Who have taken anti-inflammatory analgesics or acute and chronic diseases within one month, etc.,
* The students and related stakeholders guided by the host of this plan
* Who have the habit of smoking and drinking
* Within two weeks Have used probiotic products in powder, capsule or tablet form (including yogurt, yogurt, Yakult and other related foods)
* Food or allergic to lactic acid bacteria products
* Have had hepatobiliary and gastrointestinal surgery within 2 years (except hernia and polypectomy)

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Isometric Mid-Thigh Pull (IMTP_RFD | up to 6 weeks
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak rate of force development (RFD) parameters were recorded.
Isometric Mid-Thigh Pull (IMTP)_relative peak force | up to 6 weeks
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak rate of force development (RFD) parameters were recorded.
Wingate Anaerobic Test (WAnT)_relative peak power | up to 6 weeks
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The average relative peak power parameters were recorded.
Wingate Anaerobic Test (WAnT)_relative mean power | up to 6 weeks
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The average relative mean power parameters were recorded.
Wingate Anaerobic Test (WAnT)_fatigue index | up to 6 weeks
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The average fatigue index parameters were recorded.
The Countermovement Jump (CMJ) Test | up to 6 weeks
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. The average power (MF), were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
VO2max | up to 6 weeks
  To evaluate the maximum oxygen consumption and exercise performance, we used a treadmill (Pulsar, h/p/cosmos, Nussdorf-Traunstein, Germany) and an automatic breathing analyzer (Vmax 29c, Sensor Medics, Yorba Linda, CA, USA). In addition, a polar heart rate device was used to monitor the heart rate (HR). The speed range of the treadmill was set to 7.2 km/h and increased by 1.8 km/h every 2 min until fatigue, according to Bruce's protocol. When the breathing exchange rate (the volume ratio of carbon dioxide produced to oxygen consumed, VCO2/VO2) was higher than 1.10 and reached the maximum heart rate (maximum heart rate = 220 - age), oxygen consumption was considered to be maximum. The three highest VO2max peak were averaged to obtain the VO2max values of the individual volunteers.
Muscle composition_muscle thickness | up to 6 weeks
  Use muscular ultrasound (BenQ T3300) to scan muscle thickness
Muscle composition_fascia thickness | up to 6 weeks
  Use muscular ultrasound (BenQ T3300) to scan fascia thickness
dual-energy X-ray absorptiometry, DXA | up to 6 weeks
  A non-invasive dual-energy X-ray absorptive bone density testing room (Lunar iDXA, GE Healthcare, Chicago, IL, USA) was used for systemic body composition and bone density measurements. The subject was required to lie flat on the test bed, with their body at the center line, and their limbs within the detection range. Two different energy X-rays were used to scan the inspected part, then the scintillation detector received the X-rays that had penetrated the inspected part, and analyzed the obtained muscle mass
Body composition_body fat | up to 6 weeks
  The multi-frequency principle was applied to measure body composition by using a bioelectrical impedance analyzer (BIA) on an InBody 570 device (In-body, Seoul, South Korea). To perform the measurements, after the subjects' palms and soles were removed from the sensors, the subjects stood on the footing electrodes and held the sensing handles with two hands. During the measurements, the subjects kept their arms open and left their bodies at an angle of 30° without speaking or moving. The subjects also fasted for at least 8 h before the test. The body fat were meansure
Body composition_muscle mass | up to 6 weeks
  The multi-frequency principle was applied to measure body composition by using a bioelectrical impedance analyzer (BIA) on an InBody 570 device (In-body, Seoul, South Korea). To perform the measurements, after the subjects' palms and soles were removed from the sensors, the subjects stood on the footing electrodes and held the sensing handles with two hands. During the measurements, the subjects kept their arms open and left their bodies at an angle of 30° without speaking or moving. The subjects also fasted for at least 8 h before the test. The muscle mass were meansure
Grip strength | up to 6 weeks
  Use the armed grip machine (T.K.K.5401, Takei Scientific Instruments Co.,Ltd, Niigata, Japan) to measure, hold each of the left and right hands three times until they are weak, and record the maximum value

SECONDARY OUTCOMES:
Safety assessment - AST | up to 6 weeks
  Safety is assessed function of liver such as AST (8-38 IU/L).
Safety assessment - ALT | up to 6 weeks
  Safety is assessed function of liver such as ALT (4-44 IU/L).
Safety assessment - T-Cholesterol | up to 6 weeks
  Safety is assessed function of blood lipid such as T-Cholesterol (<200 mg/dL).
Safety assessment - Uric Acid | up to 6 weeks
  Safety is assessed function of kidney such as Uric Acid (3.4-7.6 mg/dl)
Safety assessment - BUN | up to 6 weeks
  Safety is assessed function of kidney such as Bun (6-20 mg/dl)
Safety assessment - Creatinine | up to 6 weeks
  Safety is assessed function of kidney such as Creatinine (0.6-1.3 mg/dl)
Safety assessment - Glucose | up to 6 weeks
  Safety is assessed function of Glucose (70~100 mg/dL)
Safety assessment - Triglycerides | up to 6 weeks
  Safety is assessed function of blood lipid such as Triglycerides (<150 mg/dL)
Safety assessment - LDL | up to 6 weeks
  Safety is assessed function of blood lipid such as LDL (0~140mg/dl)
Safety assessment - HDL | up to 6 weeks
  Safety is assessed function of blood lipid such as HDL (>40mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No